CLINICAL TRIAL: NCT04396288
Title: Characterization of Intra-osseous Vascular Response With Ultrasound Imaging on Healthy Volunteers
Brief Title: Ultrasound Imaging-based Measurement of Intra-osseous Vascular Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: C19-30
Record Dates: First submitted 2020-05-05; First posted 2020-05-20 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2024-03

CONDITIONS: Blood Circulation Disorder; Bone Diseases, Metabolic
MeSH Terms: conditions — Bone Diseases, Metabolic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Healthy volunteers (Experimental)
  Interventions: Device: ultrasound imaging at the forearm and at the tibia

INTERVENTIONS:
Device: ultrasound imaging at the forearm and at the tibia — ultrasound imaging will be performed at the radius bone (forearm) and at the tibia, before, during, and after a change of intraosseous blood flow

SUMMARY:
Blood circulation within bone is thought to have a key role in bone growth, in fracture healing and in the development of bone diseases like osteoporosis. Current medical imaging techniques such as conventional ultrasonography fail to detect blood circulation within bone. The investigators propose to develop a new type of ultrasonography called intraosseous functional ultrasonography that will enable the detection and the characterization of blood circulation in solid bone tissue, marrow and soft tissues surrounding bone (muscle for instance). Because most soft tissues are essentially made of water, the speed of sound in soft tissues is close to that in water and it varies only a little between different types of soft tissues. For this reason, clinical ultrasound scanners used for ultrasonography assume that the speed of sound in the human body is the same for all types of soft tissues. This assumption is reasonable in soft tissues, but it does not hold in bone because solid bone tissue is much stiffer than soft tissues. Seismologists have extensive experience in producing images of the structure of the Earth based on the analysis of elastic waves which follow the same laws of Physics as ultrasound waves. The subsurface of the Earth contains layers of solid materials and liquids, consequently it is very similar to a region of the human body containing bone and soft tissues. Therefore the investigators will first work on the adaption of time-tested seismic imaging methods to make ultrasonography of bone possible. Once a correct image of bone is obtained, the investigators will use an ultrasound scanner dedicated to research to repeat this image hundreds of times per second, very much like a slow motion video. Because blood is moving while bone is still, the intensity in the image is being slightly changed where blood is moving. Thus the analysis of these changes makes it possible to detect and characterize blood flow within bone. In this way the investigators expect to be able to detect blood flowing with a speed as low as a few millimeters per second. Finally the sensitivity of the technique to detect and characterize blood circulation in bone will be evaluated in patients at the hospital and in healthy volunteers. The success of this work will help gaining knowledge on the role of blood circulation within bone. In the long term, it may help in the diagnosis of bone diseases.

ELIGIBILITY:
Inclusion Criteria:

* be 18 years old or older
* speaks good French
* have an affiliation to a French Healthcare system (health insurance)
* sign the informed consent

Exclusion Criteria:

* bone fracture at the tibia or at the forearm less than one year ago
* injury or wound still present at the tibia or at the forearm
* pregnant women
* protected persons

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2021-09-14 (Actual); Primary Completion 2022-12-14 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Change of velocity of blood flow in cortical bone and in marrow, before, during, and after the action of an automatic blood pressure cuff at the forearm (radius bone) | Up to 10 secondes immediately before the action of an automatic blood pressure cuff, during the action of an automatic blood pressure cuff (about 20 secondes), and up to 10 secondes immediately after the action of an automatic blood pressure cuff
  Using ultrasound imaging, the velocity (mm/s) of blood circulation in cortical bone and in marrow will be assessed at the forearm (radius bone). Changes induced by the action of an automatic blood pressure cuff will be measured.
Change of direction of blood flow in cortical bone and in marrow, before, during, and after the action of an automatic blood pressure cuff at the forearm (radius bone) | Up to 10 secondes immediately before the action of an automatic blood pressure cuff, during the action of an automatic blood pressure cuff (about 20 secondes), and up to 10 secondes immediately after the action of an automatic blood pressure cuff
  Using ultrasound imaging, the direction (degree) of blood circulation in cortical bone and in marrow will be assessed at the forearm (radius bone). Changes induced by the action of an automatic blood pressure cuff will be measured.
Change of velocity of blood flow in cortical bone and in marrow at the tibia, if changing position from sitting position to supine head-down tilt position | During sitting position (up to 5 minutes), then during supine head-down tilt position (up to 5 minutes)
  Using ultrasound imaging, the velocity (mm/s) of blood circulation in cortical bone and in marrow will be assessed at the tibia. Changes induced by the change of position will be measured.
Change of direction of blood flow in cortical bone and in marrow at the tibia, if changing position from sitting position to supine head-down tilt position | During sitting position (up to 5 minutes), then during supine head-down tilt position (up to 5 minutes)
  Using ultrasound imaging, the direction (degree) of blood circulation in cortical bone and in marrow will be assessed at the tibia. Changes induced by the change of position will be measured.

SECONDARY OUTCOMES:
Repeatability of the measurement of the change of intraosseous blood circulation at the forearm under the action of an automatic blood pressure cuff | Up to 10 secondes immediately before the action of an automatic blood pressure cuff, during the action of an automatic blood pressure cuff (about 20 secondes), and up to 10 secondes immediately after the action of an automatic blood pressure cuff
  The action of the automatic blood pressure cuff will be repeated 5 times. The ultrasound transducer will be systematically removed and replaced between each repetition, in order to assess the reproducibility of the measurement.
Repeatability of the measurement of the change of intraosseous blood circulation at the tibia when changing position from sitting position to supine head-down tilt position | During sitting position (up to 5 minutes), then during supine head-down tilt position (up to 5 minutes)
  The change of position from sitting position to supine head-down tilt position will be repeated 5 times. The ultrasound transducer will be systematically removed and replaced between each repetition, in order to assess the reproducibility of the measurement.

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Radiologie polyvalente et oncologique, hôpital La Pitié-Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cloutier G, Destrempes F, Yu F, Tang A. Quantitative ultrasound imaging of soft biological tissues: a primer for radiologists and medical physicists. Insights Imaging. 2021 Sep 9;12(1):127. doi: 10.1186/s13244-021-01071-w. PMID 34499249